CLINICAL TRIAL: NCT04064008
Title: Post Market Clinical Follow-Up Study Protocol for PROFEMUR® Z Revision Femoral Stems
Status: Enrolling by invitation | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002M
Record Dates: First submitted 2019-05-18; First posted 2019-08-21 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Joint Disease
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Total Hip Arthroplasty: Single study group from a single site previously implanted with the PROFEMUR® Z Revision Femoral Stem
  Interventions: Device: PROFEMUR® Z Revision Femoral Stem

INTERVENTIONS:
Device: PROFEMUR® Z Revision Femoral Stem — Total Hip Total Hip Arthroscopy

SUMMARY:
Single center, prospective follow-up of previously implanted subjects

DETAILED DESCRIPTION:
Post Market Clinical Follow-Up Study Protocol for PROFEMUR® Z Revision Femoral Stems

ELIGIBILITY:
Inclusion Criteria:

1. Has undergone a revision for nonunion and/or hardware removal (i.e. all conditions resulting in poor quality proximal bone).
2. Subject is implanted with the PROFEMUR® Z Revision Femoral Stem at the time of their revision THA.
3. Subject is willing and able to complete required study visits or assessments.
4. Plans to be available through the 10 year postoperative follow-up visit.

Previously implanted bilateral subjects can have both THAs enrolled in the study provided:

1. the PROFEMUR Z Revision Femoral Stem was implanted in both,
2. all other aspects of the Inclusion/Exclusion Criteria are satisfied,
3. enrollment does not exceed the subject count specified in the Clinical Trial Agreement, and
4. the subject agrees to a second Informed Consent document specific to the second THA. Prospective enrollment of a previously unimplanted hip is not permitted in this study.

Exclusion Criteria:

1. Subjects currently enrolled in another clinical study which could affect the endpoints of this protocol.
2. Subject has a PROFEMUR Neck Varus/Valgus CoCr 8 Degree, Part number PHAC 1254 implanted in the enrolled THA.
3. Has or had an overt infection at the time of implantation.
4. Has or had a distant foci of infections (which may cause hematogenous spread to the implant site) at the time of implantation.
5. Has or had a rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram at the time of implantation.
6. Has or had inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable.
7. Subjects unwilling to sign the Informed Consent document.
8. Subjects with substance abuse issues.
9. Subjects with an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study.
10. Subjects who are incarcerated or have pending incarceration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Single study group from a single site previously implanted with the PROFEMUR® Z Revision Femoral Stem
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Survivorship of ProFemur Z Stem out to 10 years | 10 years.
  Kaplan-Meier survivorship at specific intervals out to 10 years follow up

SECONDARY OUTCOMES:
Revision rate of the Profemur Z stem out to 10 years | 2-5 years, 5-7 years, and 10 years.
  Cummulative revision rate at early (2-5yrs), midterm (5-7 year) and long-term (10 year) follow up.
to characterize total functional scores for subjects, as assessed by Oxford Hip Scores | 2-5 years, 5-7 years, and 10 years.
  The study will be reporting the final Oxford Hip score, which is a summary over 12 items. Each of these items is 5-level Likert scale such as from 'not at all' to 'totally'.

OTHER OUTCOMES:
to characterize total functional scores for subjects, as assessed by EQ-5D-3L scores. | 2-5 years, 5-7 years, and 10 years.
  EQ-5D-3L data will be summarized over 5 domains, namely, mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain has 3 levels: no problems, some problems, and extreme problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny Klinika, Otwock, Poland